CLINICAL TRIAL: NCT02735902
Title: Anticoagulation Alone Versus Anticoagulation and Aspirin Following Transcatheter Aortic Valve Interventions - an Open, Multicenter Randomized Controlled Trial With Two Parallel Arms (1:1)
Brief Title: Anticoagulation Alone Versus Anticoagulation and Aspirin Following Transcatheter Aortic Valve Interventions (1:1)
Acronym: AVATAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LOCAL/2016/GC-01; 2016-000352-98 (EudraCT Number)
Record Dates: First submitted 2016-04-07; First posted 2016-04-13 (Estimated); Last update posted 2024-07-24 (Actual); Status verified 2023-09

CONDITIONS: Transcatheter Aortic Valve Replacement
Keywords: antivitamins K; direct oral anti-coagulant
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vitamin K antagonist or Direct oral anticoagulant treatment (Experimental): In this group, patients will receive monotherapy via anticoagulant (AVK or DOAC) excepted rivaroxaban; this treatment given corresponds to the anticoagulant treatment the patient was receiving before surgery. A data collection book for monitoring INR values and dates for the next 12 months is given to the patient.
  Intervention: anticoagulant
  Interventions: Drug: Vitamin K antagonist or direct oral anticoagulant treatment
- vitamin K antagonist or Direct oral anticoagulant + Aspirin (Active Comparator): In this group, patients will receive combination therapy via anticoagulant (AVK or DOAC) and aspirin, whose daily dose is between 75 mg and 100 mg; the anticoagulant treatment administered corresponds to the anticoagulant treatment the patient was receiving before the procedure, monitored and adapted according to current recommendations. A data collection book for monitoring INR values and dates for the next 12 months is given to the patient.
  Intervention: anticoagulant Intervention: Aspirin
  Interventions: Drug: Vitamin K antagonist or direct oral anticoagulant treatment; Drug: Aspirin

INTERVENTIONS:
Drug: Vitamin K antagonist or direct oral anticoagulant treatment — The Vitamin K antagonist or direct oral anticoagulant treatment will be administered to obtain an International Normalized Ratio between 2 and 3 as recommended if the treatment is AVK.
  The Direct oral anticoagulant treatment : Apixaban 5 mg x2 or 2.5 mg X2, Edoxaban 30 ou 60 mg
Drug: Aspirin — Daily dose is between 75 mg and 100 mg.
  Allergic reactions to aspirin may be observed in rare cases. In case of suspicion of allergy, treatment with aspirin is stopped.
  Arms: vitamin K antagonist or Direct oral anticoagulant + Aspirin

SUMMARY:
The main objective of this study is to demonstrate that a single anticoagulant therapy is superior to a combination of anticoagulant and antiplatelet therapy on the net clinical benefit estimated at 12 months after a Transcatheter Aortic Valve Intervention (TAVI) according to BARC2 criteria (bleeding complications; Mehran et al 2011) and VARC 3 (other complications; Kappetein et al 2012)..

DETAILED DESCRIPTION:
The secondary objectives of this study are to evaluate the following at 3 months, 6 months and 12 months after TAVI in both groups:

1. Mortality (all causes).
2. Cardiovascular mortality.
3. The occurrence of myocardial infarction.
4. The occurrence of stroke.
5. The occurrence of valve thrombosis.
6. The occurrence of major bleeding (BARC ≥ 3).
7. The occurrence of minor bleeding (2 ≤ BARC <3).
8. Treatment compliance.

ELIGIBILITY:
Inclusion Criteria:

* The patient or his/her representative must have given free and informed consent and signed the consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 12 months of follow-up
* The patient underwent a successful transcutaneous implant procedure for an aortic valve
* The patient required anticoagulant treatment (AVK or DOAC) excepted rivaroxaban the day of inclusion
* The patient is stable on anticoagulant treatment

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient or his/her representative refuses to sign the consent
* It is impossible to correctly inform the patient or his/her representative
* The patient is pregnant or breastfeeding
* The patient has a contraindication (or an incompatible drug association) for a treatment used in this study
* The patient had a coronary stent for less than 12 months
* The patient does not require treatment with aspirin or any other antiplatelet agent
* The patient has a history of aspirin allergy
* High bleeding risk; such as platelets <50,000 / mm3 during screening, Hb <8.5 g / dL, history of intracranial hemorrhage or subdural hematoma, major surgery, parenchymal organ biopsy or severe trauma within 30 days before inclusion, active gastrointestinal ulcer in the last 3 months;
* History of Stroke in the last 3 months;
* Moderate or severe liver affection associated with coagulopathy
* Active infectious endocarditis
* Active tumor treated at the time of inclusion associated with expected survival less than one year
* Not following countraindications specific to the molecules used fo the patients receiving DOAC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Composite outcome of the following events: death from any cause, myocardial infarction, stroke all causes, valve thrombosis and hemorrhage ≥ 2 as defined by the VARC 3 (Valve Academic Research Consortium scale). | Month 12

SECONDARY OUTCOMES:
All cause death according to the VARC 3 criteria | month 1
All cause death according to the VARC 3 criteria | month 3
All cause death according to the VARC 3 criteria | month 6
All cause death according to the VARC 3 criteria | month 12
Death due to cardio-vascular causes according to the VARC 2 criteria | month 1
Death due to cardio-vascular causes according to the VARC 3 criteria | month 3
Death due to cardio-vascular causes according to the VARC 3 criteria | month 6
Death due to cardio-vascular causes according to the VARC 3 criteria | month 12
Myocardial infarction according to VARC 3 criteria | month 1
Myocardial infarction according to VARC 3 criteria | month 3
Myocardial infarction according to VARC 2 criteria | month 6
Myocardial infarction according to VARC 3 criteria | month 12
Stroke (all cause) according to the VARC 3 criteria | month 1
Stroke (all cause) according to the VARC 3 criteria | month 3
Stroke (all cause) according to the VARC 3 criteria | month 6
Stroke (all cause) according to the VARC 3 criteria | month 12
Valve thrombosis according to the VARC 3 criteria | Month 1
Valve thrombosis according to the VARC 3 criteria | Month 3
Valve thrombosis according to the VARC 3 criteria | Month 6
Valve thrombosis according to the VARC 3 criteria | Month 12
Major hemorrhage (BARC ≥ 3) | Month 1
Major hemorrhage (BARC ≥ 3) | Month 3
Major hemorrhage (BARC ≥ 3) | Month 6
Major hemorrhage (BARC ≥ 3) | Month 12
Minor hemorrhage (2 ≤ BARC < 3) | Month 1
Minor hemorrhage (2 ≤ BARC < 3) | Month 3
Minor hemorrhage (2 ≤ BARC < 3) | Month 6
Minor hemorrhage (2 ≤ BARC < 3) | Month 12
Observance / Modification of treatment (Questionnaire according to Girerd et al. 2001) | Month 1
Observance / Modification of treatment (Questionnaire according to Girerd et al. 2001) | Month 3
Observance / Modification of treatment (Questionnaire according to Girerd et al. 2001) | Month 6
Observance / Modification of treatment (Questionnaire according to Girerd et al. 2001) | Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Cayla, MD, PhD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (6):
- France (6):
  - CHRU de Montpellier - Hôpital Arnaud de Villeneuve, Montpellier
  - Clinique du Millénaire, Montpellier
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - Hôpital Privé les Franciscaines, Nîmes
  - Clinique Saint-Pierre, Perpignan
  - CH de Perpignan - Hôpital Saint Jean, Perpignan

REFERENCES:
- [Background] Girerd X, Radauceanu A, Achard JM, Fourcade J, Tournier B, Brillet G, Silhol F, Hanon O. [Evaluation of patient compliance among hypertensive patients treated by specialists]. Arch Mal Coeur Vaiss. 2001 Aug;94(8):839-42. French. PMID 11575214
- [Background] Kappetein AP, Head SJ, Genereux P, Piazza N, van Mieghem NM, Blackstone EH, Brott TG, Cohen DJ, Cutlip DE, van Es GA, Hahn RT, Kirtane AJ, Krucoff MW, Kodali S, Mack MJ, Mehran R, Rodes-Cabau J, Vranckx P, Webb JG, Windecker S, Serruys PW, Leon MB. Updated standardized endpoint definitions for transcatheter aortic valve implantation: the Valve Academic Research Consortium-2 consensus document. Eur Heart J. 2012 Oct;33(19):2403-18. doi: 10.1093/eurheartj/ehs255. PMID 23026477